CLINICAL TRIAL: NCT02140385
Title: Role of Preservation of Scarpa's Fascia in Abdominoplasty: a Prospective Trial
Brief Title: Role of Preservation of Scarpa's Fascia in Abdominoplasty
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 5120289
Record Dates: First submitted 2013-09-24; First posted 2014-05-16 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Abdominoplasty
MeSH Terms: interventions — Lymphoscintigraphy; Imaging, Three-Dimensional

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Abdominoplasty-Scarpa's fascia preservation (Active Comparator): Scarpa's fascia preservation Lymphoscintigraphy 3D imaging Abdominal ultrasound
  Interventions: Procedure: Abdominoplasty-Scarpa's fascia preservation; Device: Lymphoscintigraphy; Device: 3D Imaging; Device: Abdominal ultrasound
- Abdominoplasty-Scarpa's fascia ablation (Active Comparator): Scarpa's fascia ablation Lymphoscintigraphy 3D imaging Abdominal ultrasound
  Interventions: Procedure: Abdominoplasty-Scarpa's fascia ablation; Device: Lymphoscintigraphy; Device: 3D Imaging; Device: Abdominal ultrasound

INTERVENTIONS:
Procedure: Abdominoplasty-Scarpa's fascia preservation — Thicker abdominal flaps will be preserved during the surgery.
  Arms: Abdominoplasty-Scarpa's fascia preservation
Procedure: Abdominoplasty-Scarpa's fascia ablation — Thinner abdominal flaps will be preserved during surgery.
  Arms: Abdominoplasty-Scarpa's fascia ablation
Device: Lymphoscintigraphy — Post-operative lymphatic imaging will be conducted using a common radiographic medium
Device: 3D Imaging — Post-operative 3-dimensional photography will take place at a regularly scheduled clinic appointment.
Device: Abdominal ultrasound — Post-operative abdominal ultrasound will be used to determine the presence of fluid collections (seromas).

SUMMARY:
The purpose of this study is to determine whether leaving a thicker layer -which preserves the tissue called Scarpa's fascia -intact during an abdominoplasty (tummy tuck) decreases the damage to the lymphatic system.

In order to investigate the effect of leaving a thinner or slightly thicker layer intact during a tummy tuck, patients who are already planning to undergo the surgery, and who agree to participate, will be randomly assigned to two groups in a manner similar to flipping a coin. The first group will have their abdominoplasty performed with a thinner layer of abdominal wall left in place while the second group will have the surgery with a slightly thicker layer left in place. Both methods of doing a tummy tuck meet acceptable standards of care, and the aesthetic outcomes will not be negatively impacted by either of the options.

Before and after the surgery, a procedure called lymphoscintigraphy will be performed. Lymphoscintigraphy is a special type of imaging where a dye, called a radiotracer, is injected and then detected by a special camera. The pictures provided by the lymphoscintigraphy allow investigators to look at the lymphatic system, which is a small network similar to blood vessels that helps drain extra fluid. The lymphoscintigraphy will help investigators to know what method of performing the tummy tuck leaves the lymphatic system most intact.

In addition, photographs of each patient's abdomen will be taken using a special camera that allows investigators to put the photographs in the computer and compile a 3-dimensional image. Investigators will be able to look at the volume changes from swelling after the surgery using these pictures. Finally, an ultrasound will be used to help identify any seromas, or fluid collections, that may form after the surgery.

The lymphoscintigraphy, photographs and the ultrasound combined will help determine whether or not leaving a thicker or thinner layer during a tummy tuck helps preserve the fluid draining lymphatic system and whether or not that effects recovery after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* all patients ages 18-65 years who are planning to undergo elective abdominoplasty

Exclusion Criteria:

* patients with contraindications to lymphoscintigraphy
* patients with contraindications to abdominoplasty
* previous abdominal surgery or traumatic perforation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Lymphatic preservation | Two weeks post-operatively
  Lymphatic integrity will be measured pre-operatively and then again two weeks post-operatively in order to evaluate preservation of the lymphatic system.

SECONDARY OUTCOMES:
Edema | Up to six months post-operatively
  Edema will be measured by calculating volumetry using 3-dimensional photography
Seroma formation | Up to six months post-operatively
  Seroma formation will be evaluated by ultrasound at routine post-operative clinic appointments

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Hill, MD, PhD, Principal Investigator — Loma Linda University Department of Plastic Surgery
Locations (1):
- Loma Linda University Department of Plastic and Reconstructive Surgery, Loma Linda, California, United States